CLINICAL TRIAL: NCT07365969
Title: The Risk of Hysterectomy at Time of Myomectomy at Ain Shams University Hospital: A Retrospective Cohort Study.
Brief Title: Risk of Hysterectomy at Time of Myomectomy
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Maya Abdelrazek, Lecturer, Ain Shams University
Other Study IDs: FMASU MS 778/2024
Record Dates: First submitted 2026-01-17; First posted 2026-01-26 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Myomectomy; Fibroid Uterus; Hysterectomy
Keywords: hysterectomy; myomectomy; fibroid uterus
MeSH Terms: conditions — Leiomyoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient who were planned for abdomoinal myomectomy: A retrospective study on women who were candidates for abdominal myomectomy in the previous 4 years

SUMMARY:
Uterine fibroids are the commonest tumor affecting the female reproductive tract and many instances they are asymptomatic but in some women there does appear to be an association with heavy menstrual blood loss and possibly subfertility. Classically, treatment has been surgical with hysterectomy the most common approach for women who have completed their fertility and myomectomy for those who wish to conceive. The surgery can be carried out laparoscopically, vaginally and abdominally. The aim of this study is to evaluate the risk of hysterectomy at the time of myomectomy, and the associated 30-day postoperative morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Women planned for abdominal myomectomy in the previous 4 years.
* Availability of complete medical records for pre-, intra- and post-operative data.

Exclusion Criteria:

* Missing or lacking information in the patients records like preoperative assessment of the fibroid uterus.
* Absence of operative notes and relevant data in the medical files.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Women who were planned for abdominal myomectomy
Study Population: Women who were planned to undergo abdominal myomectomy in the past 4 years
Sampling Method: Probability Sample
Enrollment: 293 (Actual)
Dates: Start 2024-12-15 (Actual); Primary Completion 2025-10-15 (Actual); Study Completion 2025-10-15 (Actual)

PRIMARY OUTCOMES:
Incidence of hysterectomy at time of myomectomy. | Jan 2020- Dec 2024

SECONDARY OUTCOMES:
Characteristics of the Myomas who required hysterectomy | Jan 2020- Dec 2024
  number, site, size, Figo staging
Intraoperative complications | Jan 2020- Dec 2024
  Anesthesia complication, organ injury, blood transfusion.
Postoperative complications | Jan 2020- Dec 2024
  Anemia, hemorrhage, fever, wound infection, wound hematoma
Duration of hospital stay | Jan 2020- Dec 2024
  in days
Reoperation | Jan 2020- Dec 2024
  within 5 days of surgery
Readmission after discharge from the hospital | Jan 2020- Dec 2024
  within 14 days

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Ain Shams University, Cairo, Egypt